CLINICAL TRIAL: NCT06142591
Title: Oxycodone (10, 20 mg) in a Postoperative Dressing in Patients After Surgical Debridement of Burn Wounds. A Prospective, Double-blinded, Randomized, Controlled Trial.
Brief Title: Oxycodone (10, 20 mg) in a Postoperative Dressing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7/2023
Record Dates: First submitted 2023-10-11; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (10mg oxycodone) (Active Comparator): The burn wound was covered with a three-layer sterile dressing. The first layer was a dressing soaked in Octanisept (a solution of octenidine dihydrochloride and phenoxyethanol) with 10mg Oxycodone, the second dressing with paraffin, and the third dry dressing. Octenisept (Schulke&Mayer Poland, 1000ml) is a disinfectant liquid. The 1 gram of Octenisept contains 1 mg of octenidine dihydrochloride and 20 mg of Phenoxyethanol.
  Interventions: Drug: Oxycodone 10mg
- Group B (20mg oxycodone) (Active Comparator): The burn wound was covered with a three-layer sterile dressing. The first layer was a dressing soaked in Octanisept (a solution of octenidine dihydrochloride and phenoxyethanol) with 20mg Oxycodone, the second dressing with paraffin, and the third dry dressing. Octenisept (Schulke&Mayer Poland, 1000ml) is a disinfectant liquid. The 1 gram of Octenisept contains 1 mg of octenidine dihydrochloride and 20 mg of Phenoxyethanol.
  Interventions: Drug: Oxycodone 20mg

INTERVENTIONS:
Drug: Oxycodone 10mg — 10mg of oxycodone was added to Octenisept in the wound dressing.
  Other Names: 10mg oxycodone
  Arms: Group A (10mg oxycodone)
Drug: Oxycodone 20mg — 20mg of oxycodone was added to Octenisept in the wound dressing.
  Other Names: 20mg oxycodone
  Arms: Group B (20mg oxycodone)

SUMMARY:
The study mainly focuses on pain management using 10- or 20mg oxycodone burn wound dressing at Poznan University of Medical Sciences.

DETAILED DESCRIPTION:
Subjects were randomly assigned to one of the two treatment groups, A and B. Patients scheduled for burn surgery will sign written consent pre-operatively about procedural pain management. Group A received 10mg of oxycodone in wound dressing, while those in Group B received 20mg of oxycodone in wound dressing.

ELIGIBILITY:
Inclusion Criteria:

* adults scheduled for surgical burn treatment
* aged > 18 years
* ASA physical status 1,2 or 3

Exclusion Criteria:

* opioid abuse
* ASA physical status 4, 5

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Serum morphine concentration level [ng/ml] | Measured on the day of the procedure
  Measurement of the serum morphone concentration on the day of the procedure

SECONDARY OUTCOMES:
NRS score | Measured on the day of the procedure
  0- no pain, 10- the worst pain

OTHER OUTCOMES:
Dressing morphine concentration [mg/ml] | Measured on the day of the procedure
  Evaluation of the morphine dose

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Wieczorowska-Tobis, Prof.dr hab, Study Director — Poznań University of Medical Sciences